CLINICAL TRIAL: NCT01728324
Title: A Phase III Randomised, Partially Double-blind and Placebo-controlled Study of BI 207127 in Combination With Faldaprevir and Ribavirin for Chronic Genotype 1 Hepatitis C Infection in an Extended Population of Treatment naïve Patients That Includes Those Ineligible to Receive Peginterferon
Brief Title: Phase 3 Study of BI 207127 in Combination With Faldaprevir and Ribavirin for Treatment of Patients With Hepatitis C Infection, Including Patients Who Are Not Eligible to Receive Peginterferon: HCVerso2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241.36; 2012-003535-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-11-02; First posted 2012-11-19 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Therapeutics; Ribavirin; deleobuvir; faldaprevir

ARMS (3):
- Randomised 24-week arm (Experimental): BI 207127 in combination with FDV and RBV for 24 weeks (randomised)
  Interventions: Drug: BI 207127: 24-week treatment; Drug: Faldaprevir: 24-week treatment; Drug: RBV: 24-week treatment
- Randomised 16-week arm (Experimental): BI 207127-placebo, FDV-placebo and RBV-placebo for 8 weeks followed by BI 207127 in combination with FDV and RBV for 16 weeks (randomised)
  Interventions: Drug: BI 207127-placebo: 8-week treatment; Drug: Ribavirin-placebo: 8-week treatment; Drug: Faldaprevir-placebo: 8-week treatment; Drug: Faldaprevir: 16-week treatment; Drug: Ribavirin: 16-week treatment; Drug: BI 207127: 16-week treatment
- Allocated 24-week arm (Experimental): BI 207127 in combination with FDV and RBV for 24 weeks (allocated to patients with compensated cirrhosis)
  Interventions: Drug: Ribavirin: 24-week treatment; Drug: Faldaprevir: 24-week treatment; Drug: BI 207127: 24-week treatment

INTERVENTIONS:
Drug: BI 207127-placebo: 8-week treatment — 8 weeks of placebo treatment
  Arms: Randomised 16-week arm
Drug: Ribavirin: 24-week treatment — 24 weeks of active treatment
  Arms: Allocated 24-week arm
Drug: BI 207127: 24-week treatment — 24 weeks of active treatment
  Arms: Randomised 24-week arm
Drug: Faldaprevir: 24-week treatment — 24 weeks of active treatment
  Arms: Allocated 24-week arm
Drug: Faldaprevir: 24-week treatment — 24 weeks of active treatment
  Arms: Randomised 24-week arm
Drug: Ribavirin-placebo: 8-week treatment — 8 weeks of placebo treatment
  Arms: Randomised 16-week arm
Drug: BI 207127: 24-week treatment — 24 weeks of active treatment
  Arms: Allocated 24-week arm
Drug: Faldaprevir-placebo: 8-week treatment — 8 weeks of placebo treatment
  Arms: Randomised 16-week arm
Drug: Faldaprevir: 16-week treatment — 16 weeks of active treatment
  Arms: Randomised 16-week arm
Drug: Ribavirin: 16-week treatment — 16 weeks of active treatment
  Arms: Randomised 16-week arm
Drug: RBV: 24-week treatment — 24 weeks of active treatment
  Arms: Randomised 24-week arm
Drug: BI 207127: 16-week treatment — 16 weeks of active treatment
  Arms: Randomised 16-week arm

SUMMARY:
The aim of the study is to confirm efficacy and safety of treatment with 600 mg of BID BI 207127 in combination with 120 mg QD FDV and RBV for 16 or 24 weeks in target chronically infected HCV GT1b treatment naïve patients, including patients with compensated cirrhosis.

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C infection, diagnosed by positive anti-HCV antibodies and detected HCV RNA at screening
2. HCV infection of sub-GT1b confirmed by genotypic testing at screening.
3. HCV viral load =1,000 IU/mL at randomisation.
4. Patients who have never been previously treated with any other HCV treatment regimen.

Exclusion criteria:

1. HCV infection of mixed GT (1/2, 1/3, and 1/4) diagnosed by genotypic testing at screening.
2. HCV infection of sub-GT1a, mixed GT1a/1b, or undefined GT1.
3. Liver disease due to causes other than chronic HCV infection.
4. HIV infection.
5. Hepatitis B virus infection based on presence of HBs-Ag.
6. Confirmed or suspected active malignancy or history of malignancy within the last 5 years prior to screening.
7. History of illicit drug abuse other than cannabis or chronic alcohol abuse within 12 months prior to randomisation.
8. Subject is not willing to comply with the precautionary measures to prevent photosensitivity (avoid excessive sun exposure and use sun block on a daily basis).
9. Decompensated liver disease, or history of decompensated liver disease.
10. Clinical evidence of unstable cardiovascular disease which may further decompensate due to anemia.
11. Red blood cell disorders.
12. Body weight <40 kg or >125 kg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (109):
- United States (31):
  - 1241.36.00016 Boehringer Ingelheim Investigational Site, North Little Rock, Arkansas
  - 1241.36.00020 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1241.36.00005 Boehringer Ingelheim Investigational Site, Bakersfield, California
  - 1241.36.00009 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1241.36.00007 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1241.36.00013 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1241.36.00019 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1241.36.00034 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1241.36.00022 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 1241.36.00004 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1241.36.00006 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1241.36.00003 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 1241.36.00010 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1241.36.00024 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 1241.36.00030 Boehringer Ingelheim Investigational Site, Zephyrhills, Florida
  - 1241.36.00027 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1241.36.00033 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1241.36.00035 Boehringer Ingelheim Investigational Site, Springfield, Illinois
  - 1241.36.00001 Boehringer Ingelheim Investigational Site, Valparaiso, Indiana
  - 1241.36.00017 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1241.36.00018 Boehringer Ingelheim Investigational Site, Tupelo, Mississippi
  - 1241.36.00043 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1241.36.00032 Boehringer Ingelheim Investigational Site, Hillsborough, New Jersey
  - 1241.36.00002 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1241.36.00039 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1241.36.00031 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1241.36.00008 Boehringer Ingelheim Investigational Site, Murray, Utah
  - 1241.36.00026 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 1241.36.00044 Boehringer Ingelheim Investigational Site, Newport News, Virginia
  - 1241.36.00015 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 1241.36.00029 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Australia (9):
  - 1241.36.61005 Boehringer Ingelheim Investigational Site, Camperdown, New South Wales
  - 1241.36.61010 Boehringer Ingelheim Investigational Site, Kogarah, New South Wales
  - 1241.36.61009 Boehringer Ingelheim Investigational Site, New Lambton, New South Wales
  - 1241.36.61007 Boehringer Ingelheim Investigational Site, Randwick, New South Wales
  - 1241.36.61002 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 1241.36.61004 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1241.36.61001 Boehringer Ingelheim Investigational Site, Darlinghurst, Victoria
  - 1241.36.61008 Boehringer Ingelheim Investigational Site, Heidelberg, Victoria
  - 1241.36.61006 Boehringer Ingelheim Investigational Site, Melbourne, Victoria
- Belgium (7):
  - 1241.36.32006 Boehringer Ingelheim Investigational Site, Antwerp
  - 1241.36.32001 Boehringer Ingelheim Investigational Site, Brussels
  - 1241.36.32004 Boehringer Ingelheim Investigational Site, Edegem
  - 1241.36.32005 Boehringer Ingelheim Investigational Site, Ghent
  - 1241.36.32002 Boehringer Ingelheim Investigational Site, Leuven
  - 1241.36.32003 Boehringer Ingelheim Investigational Site, Liège
  - 1241.36.32007 Boehringer Ingelheim Investigational Site, Roeselare
- Canada (7):
  - 1241.36.01005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1241.36.01006 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1241.36.01002 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1241.36.01003 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1241.36.01001 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1241.36.01004 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1241.36.01007 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- France (8):
  - 1241.36.33001 Boehringer Ingelheim Investigational Site, Clichy
  - 1241.36.33004 Boehringer Ingelheim Investigational Site, Créteil
  - 1241.36.33002 Boehringer Ingelheim Investigational Site, Grenoble
  - 1241.36.33003 Boehringer Ingelheim Investigational Site, Paris
  - 1241.36.33008 Boehringer Ingelheim Investigational Site, Paris
  - 1241.36.33006 Boehringer Ingelheim Investigational Site, Saint-Laurent-du-Var
  - 1241.36.33005 Boehringer Ingelheim Investigational Site, Toulouse
  - 1241.36.33007 Boehringer Ingelheim Investigational Site, Villejuif
- Germany (10):
  - 1241.36.49011 Boehringer Ingelheim Investigational Site, Aachen
  - 1241.36.49001 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.36.49012 Boehringer Ingelheim Investigational Site, Dortmund
  - 1241.36.49004 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1241.36.49008 Boehringer Ingelheim Investigational Site, Erlangen
  - 1241.36.49009 Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - 1241.36.49014 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1241.36.49002 Boehringer Ingelheim Investigational Site, Hamburg
  - 1241.36.49007 Boehringer Ingelheim Investigational Site, Mainz
  - 1241.36.49013 Boehringer Ingelheim Investigational Site, Tübingen
- Greece (4):
  - 1241.36.30001 Boehringer Ingelheim Investigational Site, Athens
  - 1241.36.30002 Boehringer Ingelheim Investigational Site, Athens
  - 1241.36.30003 Boehringer Ingelheim Investigational Site, Pátrai
  - 1241.36.30004 Boehringer Ingelheim Investigational Site, Rhodes
- Italy (9):
  - 1241.36.39025 Boehringer Ingelheim Investigational Site, Antella (fi)
  - 1241.36.39023 Boehringer Ingelheim Investigational Site, Bisceglie (bat)
  - 1241.36.39021 Boehringer Ingelheim Investigational Site, Bologna
  - 1241.36.39022 Boehringer Ingelheim Investigational Site, Milan
  - 1241.36.39020 Boehringer Ingelheim Investigational Site, Palermo
  - 1241.36.39026 Boehringer Ingelheim Investigational Site, Pavia
  - 1241.36.39028 Boehringer Ingelheim Investigational Site, Pescara
  - 1241.36.39029 Boehringer Ingelheim Investigational Site, Roma
  - 1241.36.39024 Boehringer Ingelheim Investigational Site, San Giovanni Rotondo (fg)
- New Zealand (2):
  - 1241.36.64001 Boehringer Ingelheim Investigational Site, Auckland NZ
  - 1241.36.64002 Boehringer Ingelheim Investigational Site, Hamilton
- Portugal (3):
  - 1241.36.35103 Boehringer Ingelheim Investigational Site, Barreiro
  - 1241.36.35104 Boehringer Ingelheim Investigational Site, Coimbra
  - 1241.36.35101 Boehringer Ingelheim Investigational Site, Lisbon
- Spain (8):
  - 1241.36.34006 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 1241.36.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.36.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.36.34001 Boehringer Ingelheim Investigational Site, L'Hospitalet Llobregat (bcn)
  - 1241.36.34005 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.36.34008 Boehringer Ingelheim Investigational Site, Málaga
  - 1241.36.34003 Boehringer Ingelheim Investigational Site, Seville
  - 1241.36.34007 Boehringer Ingelheim Investigational Site, Vigo (Pontevedra)
- United Kingdom (11):
  - 1241.36.44003 Boehringer Ingelheim Investigational Site, Birmingham
  - 1241.36.44006 Boehringer Ingelheim Investigational Site, Edinburgh
  - 1241.36.44011 Boehringer Ingelheim Investigational Site, Hull
  - 1241.36.44013 Boehringer Ingelheim Investigational Site, Leeds
  - 1241.36.44008 Boehringer Ingelheim Investigational Site, Leicester
  - 1241.36.44001 Boehringer Ingelheim Investigational Site, London
  - 1241.36.44005 Boehringer Ingelheim Investigational Site, London
  - 1241.36.44007 Boehringer Ingelheim Investigational Site, Manchester
  - 1241.36.44010 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1241.36.44002 Boehringer Ingelheim Investigational Site, Oxford
  - 1241.36.44004 Boehringer Ingelheim Investigational Site, Plymouth

REFERENCES:
- [Derived] Sarrazin C, Castelli F, Andreone P, Buti M, Colombo M, Pol S, Calinas F, Puoti M, Olveira A, Shiffman M, Stern JO, Kukolj G, Roehrle M, Aslanyan S, Deng Q, Vinisko R, Mensa FJ, Nelson DR. HCVerso1 and 2: faldaprevir with deleobuvir (BI 207127) and ribavirin for treatment-naive patients with chronic hepatitis C virus genotype-1b infection. Clin Exp Gastroenterol. 2016 Nov 24;9:351-363. doi: 10.2147/CEG.S111116. eCollection 2016. PMID 27920566

RESULTS

PARTICIPANT FLOW:
Groups:
- 24-wk Non-cirrhotic (NC) Treatment Group: 24 weeks of treatment with 600mg twice daily (BID) deleobuvir (DBV) in combination with 120mg once a day (QD) faldaprevir (FDV) plus ribavirin (RBV) in non-cirrhotic patients.
- 16-wk Non-cirrhotic (NC) Treatment Group: Matching placebo to DBV, Matching placebo to FDV and Matching placebo to RBV for 8 weeks followed by 600mg BID DBV in combination with 120mg FDV plus RBV for 16 weeks in non-cirrhotic patients.
- 24-wk Cirrhotic (CR) Treatment Group: 24 weeks of treatment with 600mg BID deleobuvir (DBV) in combination with 120mg QD faldaprevir (FDV) plus ribavirin (RBV) in cirrhotic patients.
Period: Termination of DBV
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Started | 211 | 213 | 72
Completed | 173 | 177 | 58
Not Completed | 38 | 36 | 14
Not completed — Adverse Event | 14 | 13 | 4
Not completed — Lack of Efficacy | 14 | 12 | 8
Not completed — Withdrawal by Subject | 9 | 6 | 2
Not completed — Other than stated | 1 | 3 | 0
Not completed — Adverse Event (Placebo Period) | 0 | 1 | 0
Not completed — Protocol Violation (Placebo Period) | 0 | 1 | 0
Period: Termination of FDV
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Started | 211 | 213 | 72
Completed | 173 | 177 | 58
Not Completed | 38 | 36 | 14
Not completed — Adverse Event | 14 | 13 | 4
Not completed — Lack of Efficacy | 14 | 12 | 8
Not completed — Withdrawal by Subject | 9 | 6 | 2
Not completed — Other than stated | 1 | 3 | 0
Not completed — Adverse Event (Placebo Period) | 0 | 1 | 0
Not completed — Protocol Violation (Placebo Period) | 0 | 1 | 0
Period: Termination of RBV
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Started | 211 | 213 | 72
Completed | 172 | 176 | 57
Not Completed | 39 | 37 | 15
Not completed — Adverse Event | 15 | 16 | 5
Not completed — Lack of Efficacy | 14 | 11 | 7
Not completed — Withdrawal by Subject | 9 | 5 | 2
Not completed — Other than stated | 1 | 3 | 1
Not completed — Adverse Event (Placebo Period) | 0 | 1 | 0
Not completed — Protocol Violation (Placebo Period) | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): This analysis set includes all randomized patients who were dispensed study medication and were documented to have taken at least one dose of any study medication, either active or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group | Total
Number analyzed (Participants) | 211 | 213 | 72 | 496
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (12.5) | 50.5 (12.3) | 58.0 (8.8) | 51.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 120 | 27 | 255
  Male | 103 | 93 | 45 | 241

OUTCOME MEASURES:

1. Primary Outcome: SVR12 Rates With Historical Control
Description: Sustained Virologic Response at Week 12 post-treatment (SVR12): Plasma Hepatitis C virus (HCV) RNA level <25 IU/mL at 12 weeks after end of Treatment (EOT). SVR12, was assessed based on the observed HCV RNA result taken at least 10 weeks after treatment discontinuation. This definition was also applied to patients who discontinued treatment early: if the patient had HCV RNA undetected at least 10 weeks after stopping all treatment, they were considered a responder in the primary analysis. This is the primary analyses of the primary endpoint.
  The number of participants analyzed are actually adjusted number of participant analyzed.
Time Frame: 12 Week (post-treatment)
Population: Modified full analysis set (mFAS): included patients in the full analysis set (FAS) who received at least one dose of active treatment;
Measure: Number; unit: percentage of participants
Groups:
- 24-wk Non-cirrhotic (NC)+24-wk Cirrhotic (CR) Treatment Group: 24 weeks of treatment with 600mg BID deleobuvir (DBV) in combination with 120mg QD faldaprevir (FDV) plus ribavirin (RBV) in non-cirrhotic and cirrhotic patients.
- 16-wk Non-cirrhotic (NC)+24-wk Cirrhotic (CR) Treatment Group: This is the combination of 16 weeks of treatment with 600mg BID deleobuvir (DBV) in combination with 120mg QD faldaprevir (FDV) plus ribavirin (RBV) in non-cirrhotic patients and for 24 weeks in cirrhotic patients
Arm/Group | 24-wk Non-cirrhotic (NC)+24-wk Cirrhotic (CR) Treatment Group | 16-wk Non-cirrhotic (NC)+24-wk Cirrhotic (CR) Treatment Group
Number analyzed (Participants) | 283 | 283
percentage of participants
  PegIFN eligible | 79.95 | 76.68
  PegIFN ineligible | 88.28 | 70.78
Statistical Analysis 1: Comparison: 24-wk Non-cirrhotic (NC)+24-wk Cirrhotic (CR) Treatment Group; The proportion of patients achieving SVR12 achieved with 24 weeks of treatment with DBV/FDV/RBV in cirrhotic and non-cirrhotic patients was compared to an acceptable minimum SVR rate achieved with an approved direct acting anti-viral (DAA) in combination with PegIFN from historical data. The acceptable minimum SVR rate was an average of 71% (reference for PegIFN-eligible) and 50% (for PegIFN-ineligible patients), weighted by the sample size in each stratum; Test type: Superiority or Other; p < 0.0001, z-test; A stratified one sample z-test with 50% reference for PegIFN-ineligible and 71% for PegIFN-eligible patients was performed; Adjusted response rate = 81.10, 95% CI 2-sided [76.34 to 85.87] — The adjusted response rate was tested against the historical control SVR rate of 68% (95% Confidence Interval (CI): 76.3, 85.9)
Statistical Analysis 2: Comparison: 16-wk Non-cirrhotic (NC)+24-wk Cirrhotic (CR) Treatment Group; The proportion of patients achieving SVR12 achieved with 16 weeks of treatment of non-cirrhotic and 24 weeks of treatment of cirrhotic patients was compared to an acceptable minimum SVR rate achieved with an approved direct acting anti-viral (DAA) in combination with PegIFN from historical data. The acceptable minimum SVR rate was an average of 71% (reference for PegIFN-eligible) and 50% (for PegIFN-ineligible patients), weighted by the sample size in each stratum; Test type: Superiority or Other; p = 0.0020, z-test; [statistical method as in outcome 1, analysis 1]; Adjusted response rate = 75.89, 95% CI 2-sided [70.63 to 81.14]

2. Primary Outcome: Comparisons of SVR12 Rates Across Treatment Arms
Description: Sustained Virologic Response rates across treatment arms at Week 12 post-treatment (SVR12). This is the secondary analyses of the primary endpoint.
Time Frame: 12 Week (post-treatment)
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Number analyzed (Participants) | 211 | 213 | 72
Percentage of participants | 82.0 [76.8 to 87.2] | 75.6 [69.8 to 81.4] | 73.6 [63.4 to 83.8]
Statistical Analysis 1: Comparison: 24-wk Non-cirrhotic (NC) Treatment Group vs 16-wk Non-cirrhotic (NC) Treatment Group; Koch's stratum-adjusted Mantel Haenszel methods were used to compare durations, adjusting for stratification factors; Test type: Superiority or Other; p = 0.0532, Koch's method; Adjusted for PegIFN eligibility using Koch's method, with continuity correction; SVR12 Rates difference = 6.4, 95% CI 2-sided [-1.4 to 14.2]

3. Secondary Outcome: SVR4: Plasma HCV RNA Level <25 IU/mL at 4 Weeks After EOT.
Description: Sustained Virologic Response rates across treatment arms at Week 4 post-treatment (SVR4): Plasma HCV RNA level <25 IU/mL at 4 weeks after EOT.
Time Frame: 4 weeks (after End Of Treatment)
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Number analyzed (Participants) | 211 | 213 | 72
percentage of participants | 83.9 [78.9 to 88.8] | 80.3 [74.9 to 85.6] | 77.8 [68.2 to 87.4]
Statistical Analysis 1: Comparison: 24-wk Non-cirrhotic (NC) Treatment Group vs 16-wk Non-cirrhotic (NC) Treatment Group; Koch's stratum-adjusted Mantel Haenszel methods were used to compare durations, adjusting for stratification factors; Test type: Superiority or Other; p = 0.1671, Koch´s method; Adjusted for PegIFN eligibility using Koch´s method, with continuity correction; SVR4 Rates difference = 3.6, 95% CI 2-sided [-3.7 to 10.9]

4. Secondary Outcome: SVR24: Plasma HCV RNA Level <25 IU/mL at 24 Weeks After EOT.
Description: Sustained Virologic Response rates across treatment arms at Week 24 post-treatment (SVR24): Plasma HCV RNA level <25 IU/mL at 24 weeks after EOT.
Time Frame: 4 weeks (after End Of Treatment)
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Number analyzed (Participants) | 211 | 213 | 72
percentage of participants | 81.0 [75.8 to 86.3] | 74.2 [68.3 to 80.1] | 72.2 [61.9 to 82.6]
Statistical Analysis 1: Comparison: 24-wk Non-cirrhotic (NC) Treatment Group vs 16-wk Non-cirrhotic (NC) Treatment Group; Koch's stratum-adjusted Mantel Haenszel methods were used to compare durations, adjusting for stratification factors; Test type: Superiority or Other; p = 0.0447, Koch´s method; Adjusted for PegIFN eligibility using Koch´s method, with continuity correction; SVR24 Rates difference = -6.9, 95% CI 2-sided [-14.8 to 1.1]

5. Secondary Outcome: Prognostic Value of SVR12 Predicting SVR24
Description: The positive predictive value of SVR12 predicting SVR24 are the patients with an SVR12 (=YES) and the SVR24 was assessed.
Time Frame: 24 Week (post-treatment)
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Number analyzed (Participants) | 211 | 213 | 72
Percentage of participants | 99.0 | 99.0 | 98.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after all treatment discontinuation, upto 226 days.
Arm/Group | 24-wk Non-cirrhotic (NC) Treatment Group | 16-wk Non-cirrhotic (NC) Treatment Group | 24-wk Cirrhotic (CR) Treatment Group
Serious Adverse Events (participants affected / at risk) | 7/211 | 12/213 | 8/72
Other Adverse Events (participants affected / at risk) | 198/211 | 202/213 | 66/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 24-wk Non-cirrhotic (NC) Treatment Group (N=211) | 16-wk Non-cirrhotic (NC) Treatment Group (N=213) | 24-wk Cirrhotic (CR) Treatment Group (N=72)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 24-wk Non-cirrhotic (NC) Treatment Group (N=211) | 16-wk Non-cirrhotic (NC) Treatment Group (N=213) | 24-wk Cirrhotic (CR) Treatment Group (N=72)
Anaemia (Blood and lymphatic system disorders) | 26 | 22 | 13
Vertigo (Ear and labyrinth disorders) | 8 | 6 | 5
Ocular icterus (Eye disorders) | 27 | 16 | 2
Abdominal distension (Gastrointestinal disorders) | 6 | 8 | 7
Abdominal pain (Gastrointestinal disorders) | 16 | 16 | 4
Abdominal pain upper (Gastrointestinal disorders) | 26 | 19 | 7
Constipation (Gastrointestinal disorders) | 22 | 16 | 12
Diarrhoea (Gastrointestinal disorders) | 59 | 54 | 24
Dyspepsia (Gastrointestinal disorders) | 26 | 26 | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 5 | 4
Nausea (Gastrointestinal disorders) | 129 | 121 | 41
Vomiting (Gastrointestinal disorders) | 69 | 64 | 25
Asthenia (General disorders) | 43 | 34 | 18
Fatigue (General disorders) | 74 | 73 | 26
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 6 | 7
Jaundice (Hepatobiliary disorders) | 27 | 15 | 18
Nasopharyngitis (Infections and infestations) | 11 | 9 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 4 | 5
Sunburn (Injury, poisoning and procedural complications) | 13 | 14 | 3
Weight decreased (Investigations) | 19 | 11 | 6
Decreased appetite (Metabolism and nutrition disorders) | 34 | 27 | 14
Vitamin D deficiency (Metabolism and nutrition disorders) | 8 | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 11 | 1
Dizziness (Nervous system disorders) | 19 | 21 | 6
Dysgeusia (Nervous system disorders) | 14 | 8 | 5
Headache (Nervous system disorders) | 33 | 46 | 5
Paraesthesia (Nervous system disorders) | 15 | 17 | 3
Tremor (Nervous system disorders) | 2 | 2 | 5
Anxiety (Psychiatric disorders) | 8 | 21 | 6
Depression (Psychiatric disorders) | 16 | 9 | 4
Insomnia (Psychiatric disorders) | 35 | 25 | 10
Irritability (Psychiatric disorders) | 8 | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 20 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 11 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 12 | 5
Erythema (Skin and subcutaneous tissue disorders) | 33 | 39 | 10
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 38 | 26 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 47 | 23
Rash (Skin and subcutaneous tissue disorders) | 43 | 39 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.